CLINICAL TRIAL: NCT02651246
Title: Optional Sub-study to Intraoperative Imaging With ICG Registry
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 31915
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Lung, Prostate, Breast, Colon, Pancreatic, Renal, Bladder,Thyroid, Ovarian, Head and Neck,GI (Foregut - Esophagus),GI (Midgut) Cancer; Cancer of the Ovarian, Head and Neck,GI (Foregut - Esophagus),GI (Midgut), Sarcoma Cancer; Cancer of Neuro-onc, Parathyroid, Desmoid Tumors, Melanoma Cancer
MeSH Terms: conditions — Thyroid Diseases; Neoplasms; Desmoid Tumors | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: data collection

SUMMARY:
The primary goal of this optional sub-study is to record what tissues fluoresce in the operating room, and then to identify if these lesions are cancer when the histopathology is performed.

DETAILED DESCRIPTION:
Our objective is to collect prospective data on cancer subjects who undergo surgery and intraoperative imaging. The registry will include (but not limited to) cancer type, stage, intraoperative challenges to the surgeon, usage and results of intraoperative imaging, and recurrence surveillance.

In this protocol, subjects that receive intraoperative imaging will provide us the opportunity to record what tissues fluoresce in the operating room, and then to identify if these lesions are cancer when the histopathology is performed. Also, we will monitor any side effects or potential toxicities that may occur. This data can then be used to predict if a subject is more likely to develop a local recurrence due to missed cancer cells, metastatic lymph nodes or synchronous lesions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >= 18 years of age
* Patients presenting with any solid tumor and/or diseased tissue even benign nodules presumed to be resectable and are at risk for recurrence.
* Good operative candidate as determined by the treating physician and/or multidisciplinary team
* Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria:

* Pregnant women as determined by urinary or serum beta hCG within 72 hours of surgery
* Vulnerable patient populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients who undergo surgery and intraoperative imaging
Sampling Method: Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Number of tumor recurrence | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, MD, Ph.D, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States